CLINICAL TRIAL: NCT02333214
Title: The Effectiveness of an Exercise Program Using Video Games Associated With Conventional Physiotherapy in Physical Functioning in Frail Elderly Compared to Conventional Physiotherapy: Randomized Clinical Trial
Brief Title: Effectiveness of a Program Using Video Games Associated With Conventional Physiotherapy in Physical Functioning in Frail Elderly Compared to Conventional Physiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Monica Rodrigues Perracini, Professor as Master's and Doctoral Program in Physical Therapy, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE: 31998714.4.0000.0064
Record Dates: First submitted 2014-12-22; First posted 2015-01-07 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Frail Elderly
Keywords: Virtual Reality Therapy; Video Game; Physical Exercise; Aged; Frailty
MeSH Terms: conditions — Motor Activity; Frailty | interventions — Exergaming; Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exergame + conventional physiotherapy (Experimental): This group will be submitted to 30 minutes of conventional physiotherapy and 20 minutes of therapy using interactive games Xbox 360 Video Game and Entertainment Microsoft System with Kinect sensor, intervention twice a week for 12 weeks. Each game has three difficulty levels that can be used according to the performance of each participant. The protocol of conventional physiotherapy will be customized and will include exercises to improve strength and muscle power, flexibility, mobility, balance, and aerobic conditioning exercises. In particular cases, when necessary analgesia will be used to relive pain.
  Interventions: Other: Exergames and conventional physiotherapy
- Conventional physiotherapy (Active Comparator): The control group will receive 50 minutes of conventional physiotherapy intervention twice a week for 12 weeks. The protocol of conventional physiotherapy will be customized and will include exercises to improve strength and muscle power, flexibility, mobility, balance, and aerobic conditioning exercises. In particular cases, when necessary analgesia will be used to relive pain.
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Other: Exergames and conventional physiotherapy — The protocol of conventional physiotherapy will be customized and will include exercises to improve strength and muscle power, flexibility, mobility, balance, and aerobic conditioning exercises. In particular cases, when necessary analgesia will be used to relive pain. The progression of the exercises will be individualized according to the treatment plan established in the initial functional assessment and will be target to meet patient's improvement during treatment. Conventional physiotherapy will be conducted in pairs. In this group exercises that are best accomplished using virtual scenarios, such as dual task exercises, anticipatory adjustments exercises and inter limb coordination exercises will be performed using video games.
  Other Names: Experimental Group
  Arms: Exergame + conventional physiotherapy
Other: Conventional physiotherapy — The protocol of conventional physiotherapy will be customized and will include exercises to improve strength and muscle power, flexibility, mobility, balance, and aerobic conditioning exercises. In particular cases, when necessary analgesia will be used to relive pain. The progression of the exercises will be individualized according to the treatment plan established in the initial functional assessment and will be target to meet patient's improvement during treatment. Conventional physiotherapy will be conducted in pairs. In this group dual task exercises, anticipatory adjustments exercises and inter limb coordination exercises will be performed without the virtual environment.
  Other Names: Control Group
  Arms: Conventional physiotherapy

SUMMARY:
Frailty is a highly prevalent condition, reaching approximately 7% to 30% of older adults aged from 65 up to 80 years [2]. Although exercises seemed to be beneficial for the frail elders, there is still insufficient evidence to indicate the appropriate modality, frequency and intensity of physical exercises that were able to improve physical functioning in this population [9]. The virtual reality (VR) using interactive games (exergames) have generated broad scientific and clinical interest in recent years[10]. Studies indicate that older adults can benefit from training with exergames in improving mobility [12, 13], lower limb strength [14], cognition, particularly executive function [13], body balance [10, 15-18], reaction time [12] and may contribute indirectly to prevent falls [10, 19, 20]. But, there is still insufficient evidence to suggest that the use of exergames are superior even to other types of intervention [21-23] or in combination with conventional physiotherapy [24] The purpose of this study is to investigate the effectiveness of adding exercises using interactive videogames (exergames) in improving physical functioning on frail and pre frail older people when compared to conventional physiotherapy. A parallel randomized clinical with a 6 month follow-up period will be conducted with 82 frail community dwelling older adults. Participants randomized to the Experimental Group will be submitted to 30 minutes of conventional physiotherapy and 20 minutes of therapy using interactive games Xbox 360 Video Game and Entertainment Microsoft System with Kinect sensor.

The Control Group will receive 50 minutes of conventional physiotherapy. Both groups will receive 50 minutes of intervention twice a week for 12 weeks. Primary outcomes will be assessed by the Short Physical Performance Battery, the Usual walking speed test and Four Step Square Test in the baseline, 3 and 6 months after that.

DETAILED DESCRIPTION:
Frailty is considered a biological geriatric syndrome, characterized by a decreased resistance to stresses and functional reserve due to the cumulative decline in multiple physiological systems, with consequent increased state of vulnerability [2]. Negative health related outcomes, such as disability, recurrent hospitalization, institutionalization, falls and mortality [2-4] are associated with frailty, considered an emerging public health problem [2, 5]. Physical exercise has been recommended as an intervention strategy for the prevention and rehabilitation of the mobility-related outcome in the frail elderly whit positive impact on functional capacity and performance [8].

A functional downward spiral characterized by an impairment of several functional domains, such as strength, muscular endurance and motor-cognitive processes, ultimately leading to restricted mobility and decreased physical activity level is commonly observed in frail older people. Interventions that promote the integration of multisensory, cognitive and motor skills can be able to motivate the older people to remain more active for longer periods, despite their limitations. Exergames involve tasks in virtual environments that combine physical and cognitive demands in an attractive and challenging way. The player is encouraged to achieve goals and overcome limits during the game, providing immediate feedback in relation to their performance. The game experience can create a greater sense of self-efficacy and generate a more positive perception of personal skills, modulated by a positive environment reinforcement, consequently increasing motivation and engagement. This combination of greater sense of self-efficacy and greater motivation could provide a positive and necessary influence for most older people to overcome their limitations and create new lifestyle habits [25], decreasing disability. This study sought to investigate the effectiveness of adding exercises using interactive videogames (exergames) in improving physical functioning on frail and pre frail older people when compared to conventional physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

Community dwelling older adults without severe cognitive impairment (defined as a Mini Mental State Examination (MMSE) score adjusted according to the educational level with reference cutoff scores of: 13 points for those who are illiterate, ; 18 points for those with elementary and middle levels, and 26 points for those who have a high level 26), without any physiotherapy intervention for at least three months and classified as frail or pre-frail, according to the phenotype of frailty using Fried et al. criteria:

1. Unintentional weight loss of ≥ 5% or ≥ 4.5kg body weight in the previous year.
2. Exhaustion assessed by self-reported fatigue, indicated by two questions of the Center for Epidemiological Studies - Depression: (a) I felt that everything I did was an effort; (b) I could not get going. . Subjects answering "2" or "3" to either of these questions are categorized as frail by the exhaustion criterion.
3. Decreased grip strength (kg/force) in the dominant hand adjusted according to sex and body mass index (BMI). The cutoff for grip strength (Kg) criterion for men 2will be: BMI ≤ 24 grip strength ≤ 29; BMI 24,1 - 28 grip strength ≤ 30; BMI > 28 grip strength ≤ 32. The cutoff for grip strength (Kg) criterion for women will be 2: BMI ≤ 23 - grip strength ≤ 17; BMI 23,1 - 26 grip strength ≤ 17,3; BMI 26,1 - 29 grip strength ≤ 18; BMI > 29 grip strength ≤ 21.
4. Low level of physical activity. Participants will meet the criterion for physical inactivity if, in the last two weeks they did not perform a planned physical activity at least twice a week lasting more than 30 minutes or, if they did not perform planned or unplanned walks lasting for more than 15 minutes at least twice a week or, if they had performed any moderate or vigorous housework activity (> 2,5 METS) such as: wash or mop the floor, vacuuming, washing windows or wash the car frequently at least 1x a week for 30 minutes.
5. Slow walking speed. The time to walk a 4.6 meters path, with two meters for acceleration and two for deceleration, will be measured The velocity for each participant will be recorded. Those with a gait speed equal or less than 0.8 m/s will be considered frail.

Exclusion Criteria:

Severe visual impairment that prevents interaction with video games, if they had a localized loss of muscle strength and/or changes in postural tone that impede the execution of safe displacement movements in the standing position, without the aid of another person and, if they present chronic or acute diseases that contra-indicate therapeutic exercises.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in the Short Physical Performance Battery | baseline, immediately after the intervention (12 weeks) and at 6 months
  Three batteries of tests covering dimensions: balance, usual walking speed and sit-to-stand test, with scores ranging from zero (worst performance) to 12 points (best performance).
Change in the Usual walking speed test | baseline, immediately after the intervention (12 weeks) and at 6 months
  The test will be conducted on a flat surface with 8.6 meters free marked by black tape at intervals of two meters, 4,6 meters and two meters and the participant will be instructed to walk at their usual pace using their usual footwear.
Change in the Four Step Square Test | baseline, immediately after the intervention (12 weeks) and at 6 months
  Assessment of participants balance and their ability to carry out changes in the direction of the step forward, backward, and sideways, surpassing a low obstacle.

SECONDARY OUTCOMES:
Change in the The timed 5-step test | baseline, immediately after the intervention (12 weeks) and at 6 months
  Assessment of participants dynamic balance. During the test the participant will step forward and up and backward and down from a 10.1 cm step five times as fast as possible
Change in the Falls Efficacy Scale International (FES-I Brasil) | baseline, immediately after the intervention (12 weeks) and at 6 months
  The scale consists of 16 items that describe the activities of daily life and the participants should answer the level of concern of falling during these activities.
Change in the Dual task walking speed | baseline, immediately after the intervention (12 weeks) and at 6 months
  To assess the attentional demand during walking, we will use the test of usual walking speed in a 4.6 meters path with dual task. The participant will be asked to tell the evaluator an important fact of their past (the happiest day of his life, for example) along the way while walking.

CONTACTS AND LOCATIONS:
Overall Officials: Monica R Perracini, Phd, Principal Investigator — Universidade Cidade de Sao Paulo
Locations (1):
- Universidade Cidade de São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Abellan van Kan G, Rolland Y, Houles M, Gillette-Guyonnet S, Soto M, Vellas B. The assessment of frailty in older adults. Clin Geriatr Med. 2010 May;26(2):275-86. doi: 10.1016/j.cger.2010.02.002. PMID 20497846
- [Background] Malmstrom TK, Miller DK, Morley JE. A comparison of four frailty models. J Am Geriatr Soc. 2014 Apr;62(4):721-6. doi: 10.1111/jgs.12735. Epub 2014 Mar 17. PMID 24635726
- [Background] Rockwood K, Andrew M, Mitnitski A. A comparison of two approaches to measuring frailty in elderly people. J Gerontol A Biol Sci Med Sci. 2007 Jul;62(7):738-43. doi: 10.1093/gerona/62.7.738. PMID 17634321
- [Background] Bergman H, Ferrucci L, Guralnik J, Hogan DB, Hummel S, Karunananthan S, Wolfson C. Frailty: an emerging research and clinical paradigm--issues and controversies. J Gerontol A Biol Sci Med Sci. 2007 Jul;62(7):731-7. doi: 10.1093/gerona/62.7.731. PMID 17634320
- [Background] Studenski S, Hayes RP, Leibowitz RQ, Bode R, Lavery L, Walston J, Duncan P, Perera S. Clinical Global Impression of Change in Physical Frailty: development of a measure based on clinical judgment. J Am Geriatr Soc. 2004 Sep;52(9):1560-6. doi: 10.1111/j.1532-5415.2004.52423.x. PMID 15341562
- [Background] Abate M, Di Iorio A, Di Renzo D, Paganelli R, Saggini R, Abate G. Frailty in the elderly: the physical dimension. Eura Medicophys. 2007 Sep;43(3):407-15. Epub 2006 Nov 22. PMID 17117147
- [Background] Gine-Garriga M, Roque-Figuls M, Coll-Planas L, Sitja-Rabert M, Salva A. Physical exercise interventions for improving performance-based measures of physical function in community-dwelling, frail older adults: a systematic review and meta-analysis. Arch Phys Med Rehabil. 2014 Apr;95(4):753-769.e3. doi: 10.1016/j.apmr.2013.11.007. Epub 2013 Nov 27. PMID 24291597
- [Background] de Bruin ED, Schoene D, Pichierri G, Smith ST. Use of virtual reality technique for the training of motor control in the elderly. Some theoretical considerations. Z Gerontol Geriatr. 2010 Aug;43(4):229-34. doi: 10.1007/s00391-010-0124-7. PMID 20814798
- [Background] Levin MF. Can virtual reality offer enriched environments for rehabilitation? Expert Rev Neurother. 2011 Feb;11(2):153-5. doi: 10.1586/ern.10.201. No abstract available. PMID 21306202
- [Background] Bisson E, Contant B, Sveistrup H, Lajoie Y. Functional balance and dual-task reaction times in older adults are improved by virtual reality and biofeedback training. Cyberpsychol Behav. 2007 Feb;10(1):16-23. doi: 10.1089/cpb.2006.9997. PMID 17305444
- [Background] Maillot P, Perrot A, Hartley A. Effects of interactive physical-activity video-game training on physical and cognitive function in older adults. Psychol Aging. 2012 Sep;27(3):589-600. doi: 10.1037/a0026268. Epub 2011 Nov 28. PMID 22122605
- [Background] Jorgensen MG, Laessoe U, Hendriksen C, Nielsen OB, Aagaard P. Efficacy of Nintendo Wii training on mechanical leg muscle function and postural balance in community-dwelling older adults: a randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2013 Jul;68(7):845-52. doi: 10.1093/gerona/gls222. Epub 2012 Oct 31. PMID 23114461
- [Background] Bieryla KA, Dold NM. Feasibility of Wii Fit training to improve clinical measures of balance in older adults. Clin Interv Aging. 2013;8:775-81. doi: 10.2147/CIA.S46164. Epub 2013 Jun 24. PMID 23836967
- [Background] Pluchino A, Lee SY, Asfour S, Roos BA, Signorile JF. Pilot study comparing changes in postural control after training using a video game balance board program and 2 standard activity-based balance intervention programs. Arch Phys Med Rehabil. 2012 Jul;93(7):1138-46. doi: 10.1016/j.apmr.2012.01.023. Epub 2012 Mar 11. PMID 22414490
- [Background] Rendon AA, Lohman EB, Thorpe D, Johnson EG, Medina E, Bradley B. The effect of virtual reality gaming on dynamic balance in older adults. Age Ageing. 2012 Jul;41(4):549-52. doi: 10.1093/ageing/afs053. Epub 2012 Jun 6. PMID 22672915
- [Background] Szturm T, Betker AL, Moussavi Z, Desai A, Goodman V. Effects of an interactive computer game exercise regimen on balance impairment in frail community-dwelling older adults: a randomized controlled trial. Phys Ther. 2011 Oct;91(10):1449-62. doi: 10.2522/ptj.20090205. Epub 2011 Jul 28. PMID 21799138
- [Background] Duque G, Boersma D, Loza-Diaz G, Hassan S, Suarez H, Geisinger D, Suriyaarachchi P, Sharma A, Demontiero O. Effects of balance training using a virtual-reality system in older fallers. Clin Interv Aging. 2013;8:257-63. doi: 10.2147/CIA.S41453. Epub 2013 Feb 28. PMID 23467506
- [Background] Schoene D, Lord SR, Delbaere K, Severino C, Davies TA, Smith ST. A randomized controlled pilot study of home-based step training in older people using videogame technology. PLoS One. 2013;8(3):e57734. doi: 10.1371/journal.pone.0057734. Epub 2013 Mar 5. PMID 23472104
- [Background] Booth V, Masud T, Connell L, Bath-Hextall F. The effectiveness of virtual reality interventions in improving balance in adults with impaired balance compared with standard or no treatment: a systematic review and meta-analysis. Clin Rehabil. 2014 May;28(5):419-31. doi: 10.1177/0269215513509389. Epub 2013 Nov 4. PMID 24188913
- [Background] Miller KJ, Adair BS, Pearce AJ, Said CM, Ozanne E, Morris MM. Effectiveness and feasibility of virtual reality and gaming system use at home by older adults for enabling physical activity to improve health-related domains: a systematic review. Age Ageing. 2014 Mar;43(2):188-95. doi: 10.1093/ageing/aft194. Epub 2013 Dec 17. PMID 24351549
- [Background] van Diest M, Lamoth CJ, Stegenga J, Verkerke GJ, Postema K. Exergaming for balance training of elderly: state of the art and future developments. J Neuroeng Rehabil. 2013 Sep 25;10:101. doi: 10.1186/1743-0003-10-101. PMID 24063521
- [Background] Molina KI, Ricci NA, de Moraes SA, Perracini MR. Virtual reality using games for improving physical functioning in older adults: a systematic review. J Neuroeng Rehabil. 2014 Nov 15;11:156. doi: 10.1186/1743-0003-11-156. PMID 25399408
- [Background] Bandura A. Health promotion by social cognitive means. Health Educ Behav. 2004 Apr;31(2):143-64. doi: 10.1177/1090198104263660. PMID 15090118
- [Background] Bertolucci PH, Brucki SM, Campacci SR, Juliano Y. [The Mini-Mental State Examination in a general population: impact of educational status]. Arq Neuropsiquiatr. 1994 Mar;52(1):1-7. Portuguese. PMID 8002795
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Batistoni SS, Neri AL, Cupertino AP. [Validity of the Center for Epidemiological Studies Depression Scale among Brazilian elderly]. Rev Saude Publica. 2007 Aug;41(4):598-605. doi: 10.1590/s0034-89102007000400014. Portuguese. PMID 17589758
- [Background] Morley JE, Perry HM 3rd, Miller DK. Editorial: Something about frailty. J Gerontol A Biol Sci Med Sci. 2002 Nov;57(11):M698-704. doi: 10.1093/gerona/57.11.m698. No abstract available. PMID 12403796
- [Background] Ainsworth BE, Haskell WL, Whitt MC, Irwin ML, Swartz AM, Strath SJ, O'Brien WL, Bassett DR Jr, Schmitz KH, Emplaincourt PO, Jacobs DR Jr, Leon AS. Compendium of physical activities: an update of activity codes and MET intensities. Med Sci Sports Exerc. 2000 Sep;32(9 Suppl):S498-504. doi: 10.1097/00005768-200009001-00009. PMID 10993420
- [Background] Abellan van Kan G, Rolland Y, Andrieu S, Bauer J, Beauchet O, Bonnefoy M, Cesari M, Donini LM, Gillette Guyonnet S, Inzitari M, Nourhashemi F, Onder G, Ritz P, Salva A, Visser M, Vellas B. Gait speed at usual pace as a predictor of adverse outcomes in community-dwelling older people an International Academy on Nutrition and Aging (IANA) Task Force. J Nutr Health Aging. 2009 Dec;13(10):881-9. doi: 10.1007/s12603-009-0246-z. PMID 19924348
- [Background] Perera S, Mody SH, Woodman RC, Studenski SA. Meaningful change and responsiveness in common physical performance measures in older adults. J Am Geriatr Soc. 2006 May;54(5):743-9. doi: 10.1111/j.1532-5415.2006.00701.x. PMID 16696738
- [Background] Nevitt MC, Cummings SR, Kidd S, Black D. Risk factors for recurrent nonsyncopal falls. A prospective study. JAMA. 1989 May 12;261(18):2663-8. PMID 2709546
- [Background] Dite W, Temple VA. A clinical test of stepping and change of direction to identify multiple falling older adults. Arch Phys Med Rehabil. 2002 Nov;83(11):1566-71. doi: 10.1053/apmr.2002.35469. PMID 12422327
- [Background] Al-Yahya E, Dawes H, Smith L, Dennis A, Howells K, Cockburn J. Cognitive motor interference while walking: a systematic review and meta-analysis. Neurosci Biobehav Rev. 2011 Jan;35(3):715-28. doi: 10.1016/j.neubiorev.2010.08.008. Epub 2010 Sep 15. PMID 20833198
- [Background] Hall CD, Echt KV, Wolf SL, Rogers WA. Cognitive and motor mechanisms underlying older adults' ability to divide attention while walking. Phys Ther. 2011 Jul;91(7):1039-50. doi: 10.2522/ptj.20100114. Epub 2011 Apr 28. PMID 21527384
- [Background] Groll DL, To T, Bombardier C, Wright JG. The development of a comorbidity index with physical function as the outcome. J Clin Epidemiol. 2005 Jun;58(6):595-602. doi: 10.1016/j.jclinepi.2004.10.018. PMID 15878473
- [Background] Fillenbaum GG, Smyer MA. The development, validity, and reliability of the OARS multidimensional functional assessment questionnaire. J Gerontol. 1981 Jul;36(4):428-34. doi: 10.1093/geronj/36.4.428. PMID 7252074
- [Background] Ramos lR, Rosa TE, Oliveira ZM, Medina MC, Santos FR. [Profile of the elderly in a metropolitan area of southeastern Brazil: results of a domiciliary survey]. Rev Saude Publica. 1993 Apr;27(2):87-94. doi: 10.1590/s0034-89101993000200003. Portuguese. PMID 8278785
- [Background] Memoria CM, Yassuda MS, Nakano EY, Forlenza OV. Brief screening for mild cognitive impairment: validation of the Brazilian version of the Montreal cognitive assessment. Int J Geriatr Psychiatry. 2013 Jan;28(1):34-40. doi: 10.1002/gps.3787. Epub 2012 Feb 27. PMID 22368034
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Cruice M, Worrall L, Hickson L. Reporting on psychological well-being of older adults with chronic aphasia in the context of unaffected peers. Disabil Rehabil. 2011;33(3):219-28. doi: 10.3109/09638288.2010.503835. Epub 2010 Jul 14. PMID 20629580
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Gobbens RJ, Luijkx KG, Wijnen-Sponselee MT, Schols JM. Toward a conceptual definition of frail community dwelling older people. Nurs Outlook. 2010 Mar-Apr;58(2):76-86. doi: 10.1016/j.outlook.2009.09.005. PMID 20362776
- [Background] Miller DK, Morrison MJ, Blair SD, Miller JP, Morley JE. Predilection for frailty remedial strategies among black and white seniors. South Med J. 1998 Apr;91(4):375-80. doi: 10.1097/00007611-199804000-00013. PMID 9563432
- [Background] Chan TC, Chan F, Shea YF, Lin OY, Luk JK, Chan FH. Interactive virtual reality Wii in geriatric day hospital: a study to assess its feasibility, acceptability and efficacy. Geriatr Gerontol Int. 2012 Oct;12(4):714-21. doi: 10.1111/j.1447-0594.2012.00848.x. Epub 2012 Apr 2. PMID 22469232
- [Background] Franco JR, Jacobs K, Inzerillo C, Kluzik J. The effect of the Nintendo Wii Fit and exercise in improving balance and quality of life in community dwelling elders. Technol Health Care. 2012;20(2):95-115. doi: 10.3233/THC-2011-0661. PMID 22508022
- [Background] Hsu JK, Thibodeau R, Wong SJ, Zukiwsky D, Cecile S, Walton DM. A "Wii" bit of fun: the effects of adding Nintendo Wii((R)) Bowling to a standard exercise regimen for residents of long-term care with upper extremity dysfunction. Physiother Theory Pract. 2011 Apr;27(3):185-93. doi: 10.3109/09593985.2010.483267. Epub 2010 Aug 10. PMID 20698793
- [Background] Heuninckx S, Wenderoth N, Swinnen SP. Systems neuroplasticity in the aging brain: recruiting additional neural resources for successful motor performance in elderly persons. J Neurosci. 2008 Jan 2;28(1):91-9. doi: 10.1523/JNEUROSCI.3300-07.2008. PMID 18171926
- [Background] Seidler RD, Bernard JA, Burutolu TB, Fling BW, Gordon MT, Gwin JT, Kwak Y, Lipps DB. Motor control and aging: links to age-related brain structural, functional, and biochemical effects. Neurosci Biobehav Rev. 2010 Apr;34(5):721-33. doi: 10.1016/j.neubiorev.2009.10.005. Epub 2009 Oct 20. PMID 19850077
- [Background] Eng K, Siekierka E, Pyk P, Chevrier E, Hauser Y, Cameirao M, Holper L, Hagni K, Zimmerli L, Duff A, Schuster C, Bassetti C, Verschure P, Kiper D. Interactive visuo-motor therapy system for stroke rehabilitation. Med Biol Eng Comput. 2007 Sep;45(9):901-7. doi: 10.1007/s11517-007-0239-1. Epub 2007 Aug 9. PMID 17687578
- [Background] Freiberger E, Haberle L, Spirduso WW, Zijlstra GA. Long-term effects of three multicomponent exercise interventions on physical performance and fall-related psychological outcomes in community-dwelling older adults: a randomized controlled trial. J Am Geriatr Soc. 2012 Mar;60(3):437-46. doi: 10.1111/j.1532-5415.2011.03859.x. Epub 2012 Feb 10. PMID 22324753